#### NCT02833077

Study ID: VOLUMA-006

**Title:** A multicenter, single-blind, randomized, controlled study of the safety and effectiveness of JUVÉDERM VOLUMA® XC injectable gel for chin augmentation

Statistical Analysis Plan Date: 28 Feb 2017

#### 1. Title Page

#### STATISTICAL ANALYSIS PLAN

A multicenter, single-blind, randomized, controlled study of the safety and effectiveness of JUVÉDERM VOLUMA® XC injectable gel for chin augmentation

Draft 1.0: 2017-02-28

Study Number: VOLUMA-006

Development Phase: Pivotal

Product Name: JUVÉDERM VOLUMA XC Injectable

Study Statistician:

Sponsor: Allergan, Inc.

2525 Dupont Drive, Irvine, CA 92612

This document is the property of Allergan, Inc. and may not, in full or part, be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan, Inc.

## 2. Table of Contents

| 1. | Title | Page | | | 1 |
|---|---|---|---|---|---|
| 2. | Tabl | e of Co | ntents | | 2 |
| | 2.1 | List of | f Tables | | 3 |
| | | | 100100 | | |
| 3. | List | of Abbr | eviations | and Definition of Terms | 6 |
| 4. | | | | | |
| ₹. | | | | | |
| | 4.1 | Study | Design S | ummary | 7 |
| | | 4.1.0 | NT 1 | | |
| | 4.0 | 4.1.2 | | of Participants | |
| | 4.2 | Study | Objective | es and Endpoints | 9 |
| 5. | Stati | stical M | <b>lethodolo</b> | gy and Study Endpoints | 15 |
| | 5.1 | Statist | cical and A | Analytical Plans | 15 |
| | | 5.1.1 | Commo | n Conventions | 15 |
| | | | 5.1.1.1 | Analysis Populations | 15 |
| | | | 5.1.1.2 | Study Treatments | 15 |
| | | | 5.1.1.3 | Statistical Methodology | 15 |
| | | | 5.1.1.4 | Missing Data | |
| | | | 5.1.1.5 | Site Pooling | 16 |
| | | 5.1.2 | Demogr | aphics | 17 |
| | | | 5.1.2.1 | Analysis Populations | 17 |
| | | | 5.1.2.2 | Subject Disposition | |
| | | | 5.1.2.3 | Protocol Deviations | |
| | | | 5.1.2.4 | Demographics | 18 |
| | | | 5.1.2.5 | Baseline Characteristics | |
| | | | 5.1.2.6 | Medical History | 19 |
| | | | 5.1.2.7 | Prior and Concomitant Medications | |
| | | | 5.1.2.8 | Exposure to Study Treatment | |
| | | | 5.1.2.9 | Administration of Study Treatment | |
| | | 5.1.3 | Effectiv | eness Analyses | |
| | | | 5.1.3.1 | Primary Effectiveness Endpoint | |
| | | | 5.1.3.2 | Secondary Effectiveness Endpoint | |
| | | 5.1.4 | Safety A | Analyses | 23 |

| | | 5.1.4.1 S | Study Treatment Exposure and Compliance | 24 |
|---|---|---|---|---|
| | | 5.1.4.2 A | Adverse Events | 24 |
| | | 5.1.6 Interim An | and trans | 27 |
| | 5.2 | | nalysesSample Size | |
| | | | • | |
| _ | 5.3 | | onduct of the Study or Planned Analyses | |
| 6. | Data | Handling and Anal | lysis Conventions | 29 |
| | 6.1 | Analysis Days | | 29 |
| | | 6.2.1 Effectiven | ess | 30 |
| | | 6.2.2 Safety | | 31 |
| | 6.3 | Missing/Incomple | ete Date Conventions | 31 |
| | | 6.3.1 Missing/In | ncomplete AE Start Date | 31 |
| | | 6.3.2 Missing/In | ncomplete AE End Date | 32 |
| | 6.4 | Imputed Value Lis | sting Conventions | 32 |
| ŀ | | | | |
| 2.1 | | List of Tabl | les | |
| Tah | le 3-1 | Abbreviations | s and Definitions of Terms | 6 |
| 140 | | | | |

| Table 5-1 | Analysis Populations | 15 |
|------------|---------------------------------------------|----|
| Table 5-2 | Statistical Methodology | 15 |
| Table 5-3 | Missing Data Handling by Endpoint Type | 16 |
| Table 5-4 | Analysis Population Summaries | 17 |
| Table 5-5 | Subject Disposition Summaries | 17 |
| able 5-6 | Protocol Deviation Summary | 18 |
| able 5-7 | Demographic Summaries. | 18 |
| able 5-8 | Baseline Characteristics Summaries | 19 |
| able 5-9 | Medical History | 19 |
| able 5-10 | Medication | 19 |
| able 5-11 | Exposure to Study Treatment | 20 |
| Table 5-12 | Administration of Study Treatment | 20 |
| Table 5-13 | Effectiveness Assessments | 21 |
| able 5-14 | Effectiveness Endpoint Baseline Definitions | 21 |
| able 5-15 | Primary Effectiveness Analyses | 21 |
| able 5-16 | Secondary Effectiveness Analyses | 21 |
| Table 5-18 | AE Terms | 21 |
| Table 5-19 | AE Summaries | 21 |

| Table 5-26 | Sample Size Assumptions | 28 |
|------------|--------------------------|----|
| Table 6-1 | Analysis Day Definitions | 29 |

## 3. List of Abbreviations and Definition of Terms

Table 3-1 Abbreviations and Definitions of Terms

| Abbreviation/Term | Definition |
|-------------------|-----------------------------------------------------|
| 3D | 3-dimensional |
| ACRS | Allergan Chin Retrusion Scale |
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| CFR | Code of Federal Regulations |
| CI | Confidence Interval |
| eCRF | Electronic Case Report Form |
| EI | Evaluating Investigator |
| DFU | Directions For Use |
| FDA | Food and Drug Administration |
| GAIS | Global Aesthetic Improvement Scale |
| НА | Hyaluronic Acid |
| HIPAA | Health Insurance Portability and Accountability Act |
| IC | Informed Consent |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IRB | Institutional Review Board |
| ISO | International Organization for Standardization |
| ISR | Injection Site Response |
| ITT | Intent-to-treat |
| IWRS | Interactive Web Response System |
| mITT | modified Intent-To-Treat |
| PP | Per-Protocol |
| PT | Preferred Term |
| SADE | Serious Adverse Device Effect |
| SOC | System Organ Class |
| TI | Treating Investigator |
| UADE | Unanticipated Adverse Device Effect |
| US | United States |

#### 4. Introduction

This statistical analysis plan (SAP) details comprehensive, technical specifications of the statistical analyses of the effectiveness and safety data outlined and/or specified in the protocol of Study VOLUMA-006 (Amendment 4 version dated 2017-03-01). This SAP will be approved prior to database lock.

| 4.1 | Study Design Summary |
|-----|----------------------|



## 4.1.2 Number of Participants

Up to 224 subjects will be enrolled at up to 15 sites.

#### 4.2 Study Objectives and Endpoints

The objectives of this study are to evaluate the safety and effectiveness of JUVÉDERM VOLUMA XC injectable gel in augmentation of chin retrusion in adult subjects seeking improvement in chin volume deficit.

Each study primary objective, secondary objective, and other objectives are presented with corresponding endpoint(s) below:

Table 4-1 Study Objectives and Corresponding Endpoints

| Objectives | Endpoints |
|---|---|
| To evaluate and compare the effectiveness of JUVÉDERM VOLUMA XC injectable gel with no treatment control in augmentation of chin retrusion in adult subjects seeking improvement in chin volume deficit | <ul> <li>Primary Endpoint:</li> <li>Responder rate based on photo assessment of the Allergan Chin Retrusion Scale (ACRS) at month 6</li> <li>Secondary Endpoints:</li> <li>Change from baseline in overall scores of the Satisfaction with Chin module of the FACE-Q questionnaire at month 6</li> <li>Responder rate based on Evaluating Investigator (EI) assessment of global aesthetic improvement scale (GAIS) in the chin area at month 6</li> <li>Responder rate based on subject assessments of the GAIS in the chin area at month 6</li> </ul> |
| To evaluate the safety of JUVÉDERM VOLUMA XC injectable gel in augmentation of chin retrusion in adult subjects seeking improvement in chin volume deficit | |











#### 5. Statistical Methodology and Study Endpoints

#### 5.1 Statistical and Analytical Plans

Statistical analyses will be conducted using

#### **5.1.1** Common Conventions

#### 5.1.1.1 Analysis Populations

The analysis populations will consist of subjects as defined below:

Table 5-1 Analysis Populations

| Population | Definition | Study Treatment |
|---|---|---|
| Intent-to-Treat (ITT) | All randomized subjects | Randomized assignment |
| Modified Intent-to- | All subjects randomized to the treatment (treatment group) | Randomized assignment |
| Treat (mITT) | who receive at least 1 study treatment | |
| | All subjects randomized to the control group | |
| Per-Protocol (PP)<br>population | All mITT subjects who do not have any significant protocol deviations affecting the primary effectiveness endpoint | Randomized assignment |
| Safety | All subjects randomized to the treatment (treatment group) | Actual received |
| | who receive at least 1 study device treatment | |
| | All subjects randomized to the control group | |

Unless specified otherwise, all effectiveness analyses will be performed on the mITT population using the "as-randomized" assignment for each subject (ie, if a subject randomized to the control group is treated inadvertently at the start of the study, the assessments for that subject will nonetheless be included in the control group analysis). The ITT and PP populations will be used to perform sensitivity analyses for the primary effectiveness variable. All safety analyses will be conducted using the safety population.

### **5.1.1.2 Study Treatments**

The following treatment groups are defined for this study:

• Study Treatment: JUVÉDERM VOLUMA XC injectable gel

• Control Treatment: Delayed treatment

### 5.1.1.3 Statistical Methodology

The methodologies defined below apply as specified to individual endpoints defined in this SAP.

Table 5-2 Statistical Methodology

| Methodology | Description |
|---|---|
| Categorical counts | Number and percent of subjects in individual categories |
| | <ul> <li>Subjects with ≥ 1 qualifying event counted once per individual category</li> </ul> |
| | <ul> <li>N included = participants with non-missing value for by visit analysis</li> </ul> |
| Event descriptives | <ul> <li>Number and percentage of events in individual categories</li> </ul> |
| | <ul> <li>Events counted individually for each instance</li> </ul> |
| | <ul> <li>Percentage denominator = total number of events</li> </ul> |
| Continuous | <ul> <li>N included, mean, standard deviation (SD), median, minimum, maximum</li> </ul> |
| descriptives | <ul> <li>N included = subjects with non-missing value</li> </ul> |
| CFB descriptives | • Continuous descriptives for baseline, postbaseline, and change from baseline (CFB) |
| | values |
| | <ul> <li>N included = subjects with non-missing values at both baseline and the specified</li> </ul> |
| | postbaseline analysis visit |
| CFB Paired T | <ul> <li>Continuous descriptives for baseline, postbaseline, and CFB values</li> </ul> |
| | <ul> <li>P-values from a 2-sided paired t-test comparing baseline and postbaseline values</li> </ul> |
| | <ul> <li>N included = subjects with non-missing values at both baseline and the specified</li> </ul> |
| | postbaseline analysis visit |
| Responder | <ul> <li>Categorical descriptives for responders and nonresponders</li> </ul> |
| | <ul> <li>Include count and percent along with exact binomial 95% CI</li> </ul> |
| | <ul> <li>P-values from 2-sided Fisher's exact test</li> </ul> |
| | • N included = with non-missing values at both baseline and the specified postbaseline |
| | analysis visit |

#### 5.1.1.4 Missing Data

General missing data handling conventions are specified and summarized as follows:

Table 5-3 Missing Data Handling by Endpoint Type

| Endpoint type | Timing | Missing Data Handling |
|---|---|---|
| Responder | Month 6 (no-<br>treatment control<br>period) | <ul> <li>All subjects included (ITT population)</li> <li>Multiple imputation with 5 imputed datasets is applied to subjects with no postbaseline values using the below model:</li> <li>Month 6 ACRS = β<sub>0</sub>+β<sub>1</sub>Baseline ACRS + β<sub>2</sub>Month 1 ACRS + β<sub>3</sub>Month 3 ACRS</li> </ul> |
| | | where ACRS score is based on photo assessment. |
| Responder | Month 6 (no-<br>treatment control<br>period) | <ul> <li>All subject included (ITT population)</li> <li>Last observation carried forward (LOCF) for subjects with no postbaseline values</li> </ul> |

The above missing data handling conventions will only be used for sensitivity analysis of the primary effectiveness endpoint.

### 5.1.1.5 Site Pooling

The impact of investigational sites on the primary effectiveness analysis at Month 6 will be evaluated by including investigational site, treatment assignment, and their interaction as

predictor variables in a multivariate logistic regression analysis with response status on the ACRS as the dependent variable. Investigational sites with few enrolled subjects may be pooled with other sites based on subjects enrolled, geographical region, or other site characteristics. The interaction between site and treatment will be considered significant if the p-value of this interaction is less than 0.05.

### 5.1.2 Demographics

#### 5.1.2.1 Analysis Populations

The distribution of subjects within the analysis populations will be summarized as follows:

Table 5-4 Analysis Population Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| All Consented | Distribution of all randomized, | Screening period | Listing |
| | Randomized but Discontinued Before | | |
| | Treatment, Not Randomized (with Reason | | |
| | for Randomization Failure) | | |
| Not Randomized | List of not randomized subjects with | Screening period | Listing |
| | randomization failure reasons | | |
| ITT, mITT, PP and | Distribution in total and by treatment | After randomization | Categorical counts |
| Safety populations | group | | |

#### 5.1.2.2 Subject Disposition

Subject disposition encompasses the distribution of subjects who enter, complete, and discontinue during each specified analysis period (i.e., screening and treatment periods), along with eCRF-reported discontinuation reasons from each respective analysis period. A subject in the treatment group is considered a completer if s/he completes the month 12 visit without receiving repeat treatment or completes the month 1 visit after receiving repeat treatment. A subject in the control group is considered a completer if s/he completes the month 6 visit without receiving optional treatment or completes the month 6 visit after receiving optional treatment. Subject disposition will be summarized as follows:

Table 5-5 Subject Disposition Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Study disposition | Distribution in the randomized subjects in | Month 6 and final | Categorical counts |
| | total and by treatment group | | |

#### **5.1.2.3** Protocol Deviations

Protocol deviations will be defined in a separate document, including importance classification. Protocol deviations will be summarized as follows:

Table 5-6 Protocol Deviation Summary

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Important protocol | Important protocol deviation will be listed | _ | Categorical counts/ |
| deviations | | | Listing |

### 5.1.2.4 Demographics

Demographics will be summarized for mITT population in total and by treatment group as follows:

Table 5-7 Demographic Summaries

| Endpoint | | J | Description | Timing | Methodology |
|---|---|---|---|---|---|
| Age | Age (ye | ears) rela | tive to informed consent | Informed consent | Continuous |
| | date | | | | descriptives |
| Sex, race, and ethnicity | 0 | Sex | | Screening Period | Categorical counts |
| | | 0 | Female | | |
| | | 0 | Male | | |
| | 0 | Race | | | |
| | | 0 | White | | |
| | | 0 | Black or African | | |
| | | | American | | |
| | | 0 | Asian | | |
| | | 0 | American Indian or | | |
| | | | Alaska Native | | |
| | | 0 | Native Hawiaan or Other | | |
| | | | Pacific Islander | | |
| | • | Ethnici | ty | | |
| | | 0 | Hispanic or Latino | | |
| | | 0 | Not Hispanic or Latino | | |

#### **5.1.2.5** Baseline Characteristics

Baseline characteristics will be summarized in total and by treatment group for the mITT population as follows:

Table 5-8 Baseline Characteristics Summaries

| Endpoint | Timing | Methodology |
|---|---|---|
| • Sun exposure (hours per day) | Latest assessment prior to | Continuous descriptives |
| <ul> <li>Duration of Smoking</li> </ul> | randomization | |
| Fitzpatrick Skin Phototype | Latest assessment prior to | Categorical counts |
| o I, II, III, IV, V, VI | randomization | |
| Smoking history | | |

#### **5.1.2.6 Medical History**

Medical history, encompassing abnormalities, surgeries, and cosmetic procedures reported as occurring before the Screening Visit, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 18.1 or newer. Unique subjects who report medical history events will be presented as subject listing for the Safety Population.

Table 5-9 Medical History

| Endpoint | Timing | Methodology |
|---------------------------------------|------------------|-------------|
| Abnormalities and surgeries occurring | Screening Period | Listing |
| before the Screening Visit | | |

#### 5.1.2.7 Prior and Concomitant Medications

Medications will be coded using the World Health Organization (WHO) Drug Dictionary, version March 2014 or newer. Unique subjects who reported medications (Anatomical Therapeutic Chemical (ATC) 4 class and PT) will be presented as subject listing for the Safety Population.

Table 5-10 Medication

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Prior medications | Medications taken before the study | Screening Period | Listing |
| | treatment start date and time for the | prior to | |
| | treatment group and before randomization | treatment/randomiza | |
| | date and time for the control group, | tion | |
| | regardless of medication end date | | |
| Concomitant | Medications taken on or after the study | Control Period | Listing |
| medications during | treatment start date and time for the | | |
| control period | treatment group and after randomization | | |
| | date and time but before optional treatment | | |
| | date time (at month 6) for the control | | |

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| | group, regardless of medication end date | | |
| Concomitant | Medications taken on or after the study | Treatment Period | Listing |
| medications during | treatment start date and time for both | | |
| treatment period | control and treatment groups, regardless of | | |
| | medication start date | | |

#### **5.1.2.8 Exposure to Study Treatment**

Treatment exposure related variable will be summarized for safety population by treatment group as follows:

Table 5-11 Exposure to Study Treatment

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Volume injected | Initial, Touch-up, Combined initial and | Treament period | Continuous |
| | touch-up, Repeat | | descriptives |

### **5.1.2.9** Administration of Study Treatment

Variables related to administration of treatment will be summarized for safety population by treatment group as follows:

Table 5-12 Administration of Study Treatment

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| <ul> <li>Pretreatment</li></ul> | Initial, Touch-up, Repeat<br>(Repeat for Treatment Group<br>only) | Treatment period | Categorical counts |
| Pretreatment Anesthesia duration | Initial, Touch-up, Repeat<br>(Repeat for Treatmemt Group<br>only) | Treament period | Continuous<br>descriptives |

#### **5.1.3** Effectiveness Analyses

Effectiveness analyses will be based on the mITT Population.

The following effectiveness assessments are defined:

Table 5-13 Effectiveness Assessments

| Assessment | Description |
|---|---|
| Chin retrusion based on photo | Assessed by EI using the 5-point ACRS (see Appendix A). The EI will assess 2D |
| assessment | profile images of the left side of the chin rendered by the Canfield image analysis |
| | technician from the 3D images. |
| Chin retrusion based on live | EI's live ACRS assessment |
| assessment | |
| Global Aesthetic | Assessments by subject and EI based on 5-point GAIS (see Appendix B) |
| Improvement Scale (GAIS) | |
| Satisfaction with Chin | Assessed by subject response on the Satisfaction with Chin module of the validated |
| _module | FACE-Q questionnaire (see Appendix C) |

Baseline assessments for applicable effectiveness endpoints are defined as follows:

Table 5-2 Effectiveness Endpoint Baseline Definitions

| Endpoint | Description | Timing |
|---|---|---|
| Chin retrusion based on photo | Baseline refers to the photo evaluation by EI at | Randomization/ |
| assessment | randomization (or screening if no usable | Screening |
| | assessment is available at randomization) | |
| Chin retrusion based on live assessment | Baseline refers to the joint live evaluation by EI and TI at randomization (or screening if no usable assessment is available at randomization) | Randomization/<br>Screening |
| • Satisfaction with Chin module | Baseline refers to the evaluation at screening | Screening |

## **5.1.3.1** Primary Effectiveness Endpoint

The primary effectiveness endpoint will be met if the responder rate at month 6 for the treatment group is statistically greater than that for the control group at month 6 and the observed responder rate at month 6 for the treatment group is greater than 50%. A responder is a subject who shows clinically significant improvement, i.e.,  $\geq$  1-point decrease, on the ACRS from baseline based on EI assessment of 2D renderings of the chin profile.

The primary effectiveness analysis is summarized in Table 5-15.

Table 5-15 Primary Effectiveness Analyses

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Primary: Responder analysis | Superiority of the treatment group | Month 6 | Responder |
| based on photo ACRS | over no-treatment control group | | |
| | Responder rate of treatment group | | |
| | is greater than 50% | | |

The primary effectiveness analysis will be performed on the mITT population without any missing data imputation. Sensitivity analysis will be performed using ITT and PP populations as well as using missing data handling conventions as decribed in Section 5.1.1.1.4. Additionally, sensitivity analysis will be performed on mITT subjects with a baseline ACRS photo score of 2 or 3.

#### **5.1.3.2 Secondary Effectiveness Endpoint**

The secondary effectiveness analysis is summarized in Table 5-16.

Table 5-16 Secondary Effectiveness Analyses

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Secondary 1: Responder | Summary for treatment group | Month 6 | Categorical |
| analysis based on GAIS (by | | | |
| EI and by subject) | | | |
| Secondary 2: Satisfaction | Comparison of baseline vs. | Month 6 | CFB Paired T |
| with Chin module using | postbaseline for treatment group | | |
| overall score | using 2-sided paired t-test | | |

A responder on GAIS is a subject who shows improvement in the overall aesthetic assessment in the chin area (corresponds to a response of "Improved" or "Much Improved" on GAIS).

The secondary effectiveness analysis for Satisfaction with Chin module of the FACE-Q questionnaire will be conducted only if the primary endpoint is met. No additional multiplicity adjustment or gatekeeping multiple comparisons procedures are needed.





## 5.1.4 Safety Analyses

Safety analyses will be based on the Safety Population.

#### **5.1.4.1 Study Treatment Exposure and Compliance**

See section 5.1.1.2.8.

#### **5.1.4.2** Adverse Events

The following adverse event (AE) terms are defined:

Table 5-18 AE Terms

| Term | Description |
|---|---|
| Treatment- | Treatment group: An event that initially occurs or increases in severity on or after the treatment |
| emergent | start date. |
| Adverse Event | Control group: An event that initially occurs or increases in severity on or after randomization |
| (TEAE) | date. |

AEs and encompassing abnormalities, reported as occurring after the Screening Visit, will be coded using MedDRA version 18.1 or newer. A listing for all TEAEs in the treatment and control groups will be presented. Additionally, unique subjects reporting AEs as well as the number of events in the following AE categories will be summarized for treatment subjects, control subjects after optional treatment, and all treated subjects as follows:

Table 5-3 AE Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Overall summary | Overall summary only for the following categories: • Treatment-emergent AEs (TEAEs) • Treatment-related TEAEs • Treatment-related TEAEs at injection site • Treatment-related TEAEs not at injection site • All Serious AEs (SAE) • Treatment-related SAE • Discontinued due to TEAE | Treatment period | Categorical counts,<br>Event descriptives |
| TEAEs | <ul> <li>Overall summary and by SOC,<br/>PT and severity</li> </ul> | Treatment period | Categorical counts,<br>Event descriptives |
| Treatment-related TEAEs | <ul> <li>Overall summary and by SOC, PT and severity</li> <li>Overall summary by severity, duration, time to onset, resolution, and treatment required</li> </ul> | Treatment period | Categorical counts,<br>Event descriptives |
| SAEs | Overall summary and by PT | Treatment Period | Listing |
| AEs leading to discontinuation | Overall summary and by PT | Treatment Period | Listing |

Note: SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the treatment group. AEs for control group before and after optional treatment are summarized separately.

Time to onset for TEAEs will be computed as

AE start date - reference date + 1,

where, the reference date is initial treatment date for TEAEs occurring on or after initial treatment but before touch-up treatment and the reference date is touch-up treatment date for TEAEs occurring on or after touch-up treatment but before repeat treatment.

Duration for TEAEs will be computed as AE end date – AE start date + 1.







## 5.1.6 Interim Analyses

No interim analysis will be performed.

#### 5.2 Determination of Sample Size

The sample size assumptions and estimate are summarized as follows:

Table 5-4 Sample Size Assumptions

| Parameter | Assumption / Estimate |
|------------------------------|------------------------------------------|
| Primary endpoint | Chin retrusion assessment responder |
| Risk difference <sup>1</sup> | 40 (80% Voluma vs 40% Control) |
| SD | NA |
| α | 5% |
| Sides | 2 |
| Power | >99% |
| N per group | 120 in Voluma group, 40 in control group |
| Screen Fail Rate | 15% |
| Drop-out Rate | 15% |
| N total | 224 |

<sup>&</sup>lt;sup>1</sup> Based on literature/previous study VOLUMA-002 and relevant details.

#### 5.3 Changes in the Conduct of the Study or Planned Analyses

Prior to database lock, there were no changes in study conduct or planned analyses (except per protocol analysis) from what was described in the protocol and detailed in the SAP. No unplanned analyses were conducted, and the planned analyses were conducted following database lock.

### 6. Data Handling and Analysis Conventions

#### 6.1 Analysis Days

Treatment Day for effectiveness, and AE are defined as follows:

Table 6-1 Analysis Day Definitions

| Term | Description |
|---|---|
| Effectiveness | Treatment Group and Control Group (only the control subjects receiving optional treatment): |
| | Relative to the last treatment date (either the initial treatment, if no touch-up is performed, |
| Effectiveness Day | or the touch-up treatment) |
| Effectiveness Day | <ul> <li>Effectiveness Day = analysis date - last treatment start date + 1</li> <li>Effectiveness Day 1 = last treatment start date</li> </ul> |
| | Control (before receiving optional treatment): Relative to the randomization date |
| | <ul> <li>Effectiveness Day = analysis date -randomization date +1</li> <li>Effectiveness Day 1 = randomization date</li> </ul> |
| Safety (including AE | Treatment Group and Treated Control (i.e., only the control subjects receiving optional |
| Safata Day | treatment): |
| Safety Day | Relative to treatmentdate (initial and touch-up) |
| | Safety Day = analysis date – initial treatment date + 1 |
| | Safety Day 1 = initial treatment date |
| | Control (before receiving optional treatment): Relative to the randomization date |
| | <ul> <li>Safety Day = analysis date - randomization date +1</li> <li>Safety Day 1 = randomization date</li> </ul> |
| | Treatment Group Only: |
| | Relative to the repeat treatment date (after repeat treatment) |
| | Safety Day = analysis date – repeat treatment date + 1<br>Safety Day 1 = repeat treatment date |

### **6.2** Analysis Visit Windows

All scheduled and unscheduled visits with complete dates will be assigned visit windows and used for analysis. However, if a scheduled visit with incomplete date is available with no other visits with complete date during the visit window, then the visit with incomplete date may be used for analysis and the nominal visit will be used as the visit window (e.g., if the only assessment collected for Month 6 visit window is on a Month 6 CRF with incomplete date, then those data will be used for the Month 6 assessments).

If there are multiple visits occurring within a single visit window with relevant data, the visit closest to the target day will be used in the analysis of the corresponding visit windows. If 2

visits are equal distance to the target day and are the same type of visit, then the later visit will be used.

Analysis visit windows for effectiveness endpoints and safety are defined as follows:

#### **6.2.1** Effectiveness

The analysis visit windows for effectiveness endpoints are defined as follows:





#### **6.2.2** Safety

No analysis visit windows are required for TEAEs . Analysis visit windows will only be used for summarizing . For the treatment group, refer to table 6.2 for analysis visit windows . For the control group in the control period (i.e., no treatment period) refer to table 6.3 and for the control group in the treatment period refer to table 6.2.

### **6.3** Missing/Incomplete Date Conventions

#### 6.3.1 Missing/Incomplete AE Start Date

Imputation of dates with missing day and/or month is only applied to TEAEs. If adequate information is available, no imputation is needed. TEAE start dates with missing day or month will be imputed as following:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan or the initial treatment date if they have the same year, whichever is later (because TEAE onset is not expected prior to administration of study treatment)
- If day is missing but the month and year are available, then the imputed day will be the first day of the month or the initial injection date if they have the same month and year, whichever is later

#### 6.3.2 Missing/Incomplete AE End Date

Imputation of dates with missing day and/or month is only applied to TEAEs. If adequate information is available, no imputation is needed. TEAE end dates with missing day or month will be imputed as following:

• If day and month are missing but year is available, then the imputed day and month will be 31 Dec or the study exitdate if they have the same year, whichever is earlier

If day is missing but the month and year are available, then the imputed day will be the last day of the month or the study exit date if they have the same month and year, whichever is earlier

#### **6.4** Imputed Value Listing Conventions

In general, listings will present the actual partial or missing values rather than the imputed values that may be used in endpoint derivation. In instances where imputed values will be presented, imputed values will be flagged. Actual rules will be fully defined in the table, figure, and data listing specification document.

### Appendix A: Allergan Chin Retrusion Scale

Table 1: Allergan Chin Retrusion Scale (ACRS)

| Score | Grade | Description |
|---|---|---|
| 0 | None | No chin retrusion; Chin midpoint* at or in front of the lower vermilion |
| | | border vertical line |
| 1 | Minimal | Minimal chin retrusion; Chin midpoint* is between the labiomental sulcus |
| | | vertical line and lower vermilion border vertical line |
| 2 | Moderate | Moderate chin retrusion; Chin midpoint* at labiomental sulcus vertical line |
| 3 | Severe | Sever chin retrusion; Chin midpoint* slightly behind labiomental sulcus |
| | | vertical line |
| 4 | Extreme | Extreme chin retrusion*; Chin midpoint significantly behind labiomental |
| | | sulcus vertical line |

<sup>\*</sup> Chin midpoint: the midpoint between the labiomental sulcus and the inferior point of the chin

Figure 1: Lines Used in the ACRS Descriptiors











# **ALLERGAN**

Statistical Analysis Plan

